CLINICAL TRIAL: NCT07196293
Title: A Comparison Between Protemp and Flowable Light Cure Composite Material for Creating Optimal Gingival Emergence Profile and Evaluation of Peri-implant Soft Tissue; an In-vivo Study
Brief Title: A Comparison Between Protemp and Flowable Light Cure Composite Material for Creating Optimal Gingival Emergence Profile Around Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amrita Institute of Medical Sciences & Research Center (Other)
Responsible Party: Principal Investigator, Bhavin Milind Patil, Principal Investigator, Amrita Institute of Medical Sciences & Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECASM-AIMS-2023-356
Record Dates: First submitted 2025-09-14; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Customized Healing Abutment; Dental Implant; Composite Resin; Peri-Implant Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard titanium healing abutment (No Intervention): standard titanium healing abutments used
- customized healing abutment - bulk-fill flowable composite (Active Comparator)
  Interventions: Procedure: Customized Healing Abutment - bulk fill composite
- customized healing abutment - Protemp 4 (Bis-Acryl composite) (Active Comparator)
  Interventions: Procedure: customized healing abutments - Bis acryl composite materials

INTERVENTIONS:
Procedure: Customized Healing Abutment - bulk fill composite — instead of standard healing abutments , customization was done using bulk fill composite
  Arms: customized healing abutment - bulk-fill flowable composite
Procedure: customized healing abutments - Bis acryl composite materials — customized healing abutments with bis acryl composite material was used instead of standard healing abutments
  Arms: customized healing abutment - Protemp 4 (Bis-Acryl composite)

SUMMARY:
The study focuses on the critical role of the gingival emergence profile in the success of dental implants, emphasizing its importance for both peri-implant health and esthetics. The research aims to evaluate and compare the effectiveness of two common, cost-effective dental materials-light-cure composite and Protemp (a bis-acryl composite resin)-for fabricating customized healing abutments. By assessing the peri-implant tissue response to these materials, the study seeks to determine which is more suitable for creating an optimal, natural-looking soft tissue contour, thereby providing dentists with a practical and reliable alternative to more expensive options like PEEK.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Edentulous spaces to be replaced with implant-supported single crowns.
* Antagonistic natural tooth present and sound (sound periodontium) (Stable occlusion and opposing dentition)
* Good general periodontal health
* Good general health.
* Willing to participate in the study and able to sign informed consent. (Ability to attend all follow-up appointments.)

Exclusion Criteria:

* Untreated caries or periapical lesions in the opposing natural antagonistic tooth.
* Active periodontal disease.
* major active systemic disease affecting soft tissue healing
* Multiple implant supported restorations already present.
* Long edentulous spaces.
* Complete edentulous cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Gingival Index (GI) | T1: Immediately after the placement of the final prosthesis. T2: At the one-month follow-up appointment.
  Gingival Index (GI): This index is used to evaluate inflammation of the gums around the implant.
  Scale: 0 to 3.
  Interpretation: A higher score indicates a worse outcome, signifying greater gingival inflammation.
Probing depth (PI) | T1: Immediately after the placement of the final prosthesis. T2: At the one-month follow-up appointment.
  Probing Depth (PD): This is a direct clinical measurement, not a scored scale, taken in millimeters at six points around the implant.
  Interpretation: Deeper measurements are generally associated with less healthy peri-implant tissue. Therefore, a lower value indicates a better clinical outcome.
Pink Esthetic Score (PES) | T1: Immediately after the placement of the final prosthesis. T2: At the one-month follow-up appointment.
  Pink Esthetic Score (PES): This score is used to assess the aesthetic quality of the soft tissue surrounding the implant restoration.
  Scale: 0 to 14.
  Interpretation: A higher score indicates a better and more aesthetically pleasing outcome.
Pain Numeric Scale | T1: Immediately after the placement of the final prosthesis. T2: At the one-month follow-up appointment.
  Pain Numeric Rating Scale (NRS): This scale measures the patient's subjective experience of pain during the insertion of the final prosthesis.
  Scale: 0 ("no pain") to 10 ("worst pain imaginable").
  Interpretation: A higher score indicates a worse outcome, representing more severe pain.

SECONDARY OUTCOMES:
Plaque Index (PI) | T2: At the one-month follow-up appointment.
  Plaque Index (PI): This index is used to quantify the amount of dental plaque present on the implant restoration.
  Scale: 0 to 3.
  Interpretation: A higher score indicates a worse outcome, corresponding to a greater accumulation of plaque.

CONTACTS AND LOCATIONS:
Locations (1):
- Amrita School Of Dentistry, Kochi, Kerala, India